CLINICAL TRIAL: NCT00680992
Title: An Open-label, Multi-center, Phase 2 Study of Denosumab in Subjects With Giant Cell Tumor of Bone
Brief Title: Study of Denosumab in Subjects With Giant Cell Tumor of Bone
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20062004
Record Dates: First submitted 2008-05-15; First posted 2008-05-20 (Estimated); Results first posted 2018-12-10 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Cancer; Giant Cell Tumors; Giant Cell Tumor of Bone; Benign Giant Cell Tumors
Keywords: Giant Cell Tumor of Bone
MeSH Terms: conditions — Neoplasms; Giant Cell Tumors; Giant Cell Tumor of Bone | interventions — Denosumab

ARMS (1):
- Denosumab (Experimental): 120 mg administered subcutaneously (SC) every 4 weeks (Q4W) with a loading dose of 120 mg SC on study days 8 and 15.
  Interventions: Drug: Denosumab

INTERVENTIONS:
Drug: Denosumab — 120 mg administered subcutaneously (SC) every 4 weeks (Q4W) with a loading dose of 120 mg SC on study days 8 and 15.
  Other Names: AMG 162, Immunoglobulin G2 human monoclonal antibody to RANK ligand

SUMMARY:
To determine how safe denosumab is in treating subjects with giant cell tumor of bone (GCTB)

DETAILED DESCRIPTION:
To determine how safe denosumab is in treating subjects with GCTB

ELIGIBILITY:
Inclusion criteria:

* Pathologically confirmed GCTB within 1 year before study enrollment
* Measurable evidence of active disease within 1 year before study enrollment
* Subjects with surgically unsalvageable disease (eg, sacral, spinal GCTB, or multiple lesions including pulmonary metastases) OR subjects whose planned surgery includes joint resection, limb amputation, hemipelvectomy or surgical procedure resulting in severe morbidity
* Karnofsky performance status equal or greater than 50% (ie, Eastern Cooperative Oncology Group status 0, 1, or 2)
* Adults or skeletally mature adolescents (ie, radiographic evidence of at least 1 mature long bone [eg, humerus with closed growth epiphyseal plate]) equal or greater than 12 years of age
* Skeletally mature adolescents must weigh at least 45 kg
* Before any study-specific procedure is performed, the appropriate written informed consent must be obtained

Exclusion criteria:

* Currently receiving other GCTB specific treatment (eg, radiation, chemotherapy, or embolization)
* Concurrent bisphosphonate treatment
* Known or suspected current diagnosis of underlying malignancy including high grade sarcoma, osteosarcoma, fibrosarcoma, malignant giant cell sarcoma
* Known or suspected current diagnosis of non GCTB giant cell-rich tumors
* Known or suspected current diagnosis of brown cell tumor of bone or Paget's disease
* Known diagnosis of second malignancy within the past 5 years (subjects with definitively treated basal cell carcinoma and cervical carcinoma in situ are permitted)
* Prior history or current evidence of osteonecrosis/osteomyelitis of the jaw
* Active dental or jaw condition which requires oral surgery, including tooth extraction
* Non-healed dental/oral surgery
* Planned invasive dental procedure for the course of the study
* Subject currently is enrolled in or has not yet completed at least 30 days since ending other investigational device or drug study(s), or subject is receiving other investigational agent(s)
* Subject has known sensitivity to any of the products to be administered during dosing
* Unstable systemic disease including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, or myocardial infarction within 6 months before enrollment
* Subject is pregnant or breast feeding, or planning to become pregnant within 5 months after the end of treatment
* Female subject of child bearing potential is not willing to use two methods of highly effective contraception during treatment and for 5 months after the end of treatment
* Subject has any kind of disorder that compromises the ability of the subject to give written informed consent and/or to comply with study procedures

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 535 (Actual)
Dates: Start 2008-09-09 (Actual); Primary Completion 2018-05-17 (Actual); Study Completion 2018-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (31):
- United States (10):
  - Research Site, Santa Monica, California
  - Research Site, Stanford, California
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Gainesville, Florida
  - Research Site, Boston, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, New York, New York
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Greenville, South Carolina
- Australia (4):
  - Research Site, Camperdown, New South Wales
  - Research Site, Woolloongabba, Queensland
  - Research Site, East Melbourne, Victoria
  - Research Site, Nedlands, Western Australia
- Research Site, Vienna, Austria
- Canada (2):
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- France (3):
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Villejuif
- Germany (2):
  - Research Site, Bad Saarow
  - Research Site, Stuttgart
- Italy (2):
  - Research Site, Bologna
  - Research Site, Milan
- Research Site, Leiden, Netherlands
- Research Site, Warsaw, Poland
- Spain (3):
  - Research Site, Palma de Mallorca, Balearic Islands
  - Research Site, Barcelona, Catalonia
  - Research Site, Valencia, Valencia
- Research Site, Lund, Sweden
- Research Site, Birmingham, United Kingdom

REFERENCES:
- [Background] Chawla S, Henshaw R, Seeger L, Choy E, Blay JY, Ferrari S, Kroep J, Grimer R, Reichardt P, Rutkowski P, Schuetze S, Skubitz K, Staddon A, Thomas D, Qian Y, Jacobs I. Safety and efficacy of denosumab for adults and skeletally mature adolescents with giant cell tumour of bone: interim analysis of an open-label, parallel-group, phase 2 study. Lancet Oncol. 2013 Aug;14(9):901-8. doi: 10.1016/S1470-2045(13)70277-8. Epub 2013 Jul 16. PMID 23867211
- [Background] Martin-Broto J, Cleeland CS, Glare PA, Engellau J, Skubitz KM, Blum RH, Ganjoo KN, Staddon A, Dominkus M, Feng A, Qian Y, Braun A, Jacobs I, Chung K, Atchison C. Effects of denosumab on pain and analgesic use in giant cell tumor of bone: interim results from a phase II study. Acta Oncol. 2014 Sep;53(9):1173-9. doi: 10.3109/0284186X.2014.910313. Epub 2014 May 19. PMID 24834795
- [Background] Rutkowski P, Ferrari S, Grimer RJ, Stalley PD, Dijkstra SP, Pienkowski A, Vaz G, Wunder JS, Seeger LL, Feng A, Roberts ZJ, Bach BA. Surgical downstaging in an open-label phase II trial of denosumab in patients with giant cell tumor of bone. Ann Surg Oncol. 2015 Sep;22(9):2860-8. doi: 10.1245/s10434-015-4634-9. Epub 2015 Jun 2. PMID 26033180
- [Background] Chawla S, Blay JY, Rutkowski P, Le Cesne A, Reichardt P, Gelderblom H, Grimer RJ, Choy E, Skubitz K, Seeger L, Schuetze SM, Henshaw R, Dai T, Jandial D, Palmerini E. Denosumab in patients with giant-cell tumour of bone: a multicentre, open-label, phase 2 study. Lancet Oncol. 2019 Dec;20(12):1719-1729. doi: 10.1016/S1470-2045(19)30663-1. Epub 2019 Nov 6. PMID 31704134
- [Background] Engellau J, Seeger L, Grimer R, Henshaw R, Gelderblom H, Choy E, Chawla S, Reichardt P, O'Neal M, Feng A, Jacobs I, Roberts ZJ, Braun A, Bach BA. Assessment of denosumab treatment effects and imaging response in patients with giant cell tumor of bone. World J Surg Oncol. 2018 Sep 19;16(1):191. doi: 10.1186/s12957-018-1478-3. PMID 30231890
- [Background] Bukata SV, Blay JY, Rutkowski P, Skubitz K, Henshaw R, Seeger L, Dai T, Jandial D, Chawla S. Denosumab Treatment for Giant Cell Tumor of the Spine Including the Sacrum. Spine (Phila Pa 1976). 2021 Mar 1;46(5):277-284. doi: 10.1097/BRS.0000000000003728. PMID 33038190
- [Derived] Palmerini E, Seeger LL, Gambarotti M, Righi A, Reichardt P, Bukata S, Blay JY, Dai T, Jandial D, Picci P. Malignancy in giant cell tumor of bone: analysis of an open-label phase 2 study of denosumab. BMC Cancer. 2021 Jan 22;21(1):89. doi: 10.1186/s12885-020-07739-8. PMID 33482769
- [Derived] Uday S, Gaston CL, Rogers L, Parry M, Joffe J, Pearson J, Sutton D, Grimer R, Hogler W. Osteonecrosis of the Jaw and Rebound Hypercalcemia in Young People Treated With Denosumab for Giant Cell Tumor of Bone. J Clin Endocrinol Metab. 2018 Feb 1;103(2):596-603. doi: 10.1210/jc.2017-02025. PMID 29211870
- [Derived] van der Heijden L, van de Sande MA, Hogendoorn PC, Gelderblom H, Dijkstra PD. Neoadjuvant denosumab for extensive giant cell tumor in os ischium: a case report. Acta Orthop. 2015 Jun;86(3):393-5. doi: 10.3109/17453674.2014.1002345. Epub 2015 Feb 14. No abstract available. PMID 25684041
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adults and skeletally mature adolescents (≥12 years of age) were enrolled in this open-label single-arm study. The study was conducted at 30 centers in North America, Europe, and Australia from 09 Sep 2008 to study completion on 17 May 2018. The planned study duration for each participant was at least 60 months (following protocol amendment 7).
Pre-assignment Details: 3 participants from study 20040215 (NCT00396279) were enrolled directly into safety follow-up phase without retreatment. They were excluded from all defined analysis sets and results are reported for the 532 participants enrolled into the treatment phase. Non-completion reasons are summarized for the on-study period (ie, initial treatment phase).
Groups:
- Cohort 1 (Denosumab 120 mg Q4W): Participants with surgically unsalvageable disease (eg, sacral, spinal giant cell tumor of bone (GCTB), or multiple lesions including pulmonary metastases) were enrolled into cohort 1 and received denosumab 120 milligrams (mg) subcutaneously (SC) once every 4 weeks (Q4W), starting on study day 1, plus loading doses of 120 mg SC on days 8 and 15 in the first month of treatment.
- Cohort 2 (Denosumab 120 mg Q4W): Participants with surgically salvageable disease whose planned initial on-study surgery was associated with severe morbidity (eg, joint resection, limb amputation, or hemipelvectomy) were enrolled into cohort 2 and received denosumab 120 mg SC Q4W, starting on study day 1, plus loading doses of 120 mg SC on days 8 and 15 in the first month of treatment.
- Cohort 3 (Denosumab 120 mg Q4W): Participants who participated in study 20040215 and were eligible to enroll in the current study (20062004) for continuation of treatment were enrolled into cohort 3 and received denosumab 120 mg SC Q4W, starting on study day 1. Participants in cohort 3 did not receive loading doses of denosumab on days 8 and 15 in the first month of treatment.
Period: Overall Study
Arm/Group | Cohort 1 (Denosumab 120 mg Q4W) | Cohort 2 (Denosumab 120 mg Q4W) | Cohort 3 (Denosumab 120 mg Q4W)
Started | 268 | 252 | 12
Safety Analysis Set (Received ≥1 dose of denosumab) | 265 | 249 | 12
Efficacy Analysis Set (Eligible for study and received ≥1 dose of denosumab) | 260 | 242 | 11
Completed (Completed the initial treatment phase) | 0 | 0 | 0
Not Completed | 268 | 252 | 12
Not completed — Complete Resection (as per protocol) | 25 | 121 | 0
Not completed — Administrative Decision | 83 | 42 | 5
Not completed — End of Trial | 32 | 12 | 3
Not completed — Withdrawal by Subject | 33 | 11 | 1
Not completed — Adverse Event | 21 | 19 | 1
Not completed — Other | 19 | 14 | 1
Not completed — Disease Progression | 21 | 9 | 0
Not completed — Lost to Follow-up | 12 | 14 | 0
Not completed — Noncompliance | 4 | 6 | 0
Not completed — Requirement for Alternative Therapy | 8 | 2 | 0
Not completed — Pregnancy | 5 | 0 | 1
Not completed — Death | 5 | 1 | 0
Not completed — Ineligibility Determined | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The overall baseline population consisted of the 532 participants enrolled into the treatment phase of the study.
Groups:
- Cohort 1 (Denosumab 120 mg Q4W): Participants with surgically unsalvageable disease (eg, sacral, spinal GCTB, or multiple lesions including pulmonary metastases) were enrolled into cohort 1 and received denosumab 120 mg SC once Q4W, starting on study day 1, plus loading doses of 120 mg SC on days 8 and 15 in the first month of treatment.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (Denosumab 120 mg Q4W) | Cohort 2 (Denosumab 120 mg Q4W) | Cohort 3 (Denosumab 120 mg Q4W) | Total
Number analyzed (Participants) | 268 | 252 | 12 | 532
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14 | 14 | 0 | 28
  Between 18 and 65 years | 238 | 231 | 12 | 481
  >=65 years | 16 | 7 | 0 | 23
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.4 (14.6) | 35.1 (13.5) | 36.1 (14.9) | 35.8 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 154 | 142 | 5 | 301
  Male | 114 | 110 | 7 | 231
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White or Caucasian | 221 | 208 | 11 | 440
  Black or African American | 18 | 12 | 0 | 30
  Hispanic or Latino | 13 | 13 | 1 | 27
  Asian | 11 | 14 | 0 | 25
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Other | 5 | 4 | 0 | 9
GCTB Disease Type [Number; unit: Participants]
  Primary resectable | 0 | 167 | 0 | 167
  Primary unresectable | 93 | 0 | 2 | 95
  Recurrent resectable | 0 | 85 | 0 | 85
  Recurrent unresectable | 175 | 0 | 10 | 185

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: AE defined as any untoward medical occurrence in a clinical trial participant. Serious AE defined as AE that is fatal, life threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or other significant medical hazard. Severity of AEs assessed according to Common Terminology Criteria for Adverse Events (CTCAE, v3.0) based on the general guideline: Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe; Grade 4: Life-threatening or disabling; Grade 5: Death related to AE. Investigator assessed AEs for relatedness to study drug. Results are presented for treatment-emergent events (TEAEs) and included all AEs occurring from first dose in initial treatment phase to end of initial treatment phase (or for participants entering retreatment, from first dose in initial treatment phase until end of retreatment phase).
Time Frame: From first dose of study drug up to last study visit for treatment-emergent period (a maximum of approximately 111 months).
Population: The safety analysis set included all enrolled participants who received at least one dose of denosumab on the study.
Measure: Number; unit: Participants
Arm/Group | Cohort 1 (Denosumab 120 mg Q4W) | Cohort 2 (Denosumab 120 mg Q4W) | Cohort 3 (Denosumab 120 mg Q4W)
Number analyzed (Participants) | 265 | 249 | 12
Participants
  Any TEAE | 260 | 231 | 12
  Serious TEAE | 98 | 39 | 5
  Fatal TEAE | 8 | 3 | 0
  TEAE leading to treatment phase discontinuation | 27 | 24 | 1
  TEAE leading to study drug discontinuation | 27 | 23 | 1
  CTCAE Grade 3, 4, or 5 | 121 | 59 | 6
  Any TEAE related to study drug | 184 | 136 | 9

2. Primary Outcome: Number of Participants Who Experienced the Maximum Toxicity Grade (CTCAE Grade ≥ 3) in the Indicated Clinical Chemistry Parameters
Description: Serum samples for clinical chemistry were collected on study day 1 (baseline), day 15, week 5 and each study visit Q4W thereafter until last study visit for the on-study period (ie, until end of initial treatment phase). The parameters included albumin, calcium (albumin-adjusted), creatinine, magnesium and phosphate. Results are presented for number of participants who experienced the maximum toxicity grade for each of these clinical parameters. The maximum toxicity grade experienced by each participant was based on CTCAE, v3.0, and are summarized for Grade 3 and 4. Increases and decreases in relationship to the normal parameter ranges are indicated as 'Above' and 'Below' respectively.
Time Frame: Baseline (day 1) up to last study visit for initial treatment phase (median duration approximately 30 months up to a maximum of approximately 109 months).
Population: The safety analysis set included all enrolled participants who received at least one dose of denosumab on the study.
Measure: Number; unit: Participants
Arm/Group | Cohort 1 (Denosumab 120 mg Q4W) | Cohort 2 (Denosumab 120 mg Q4W) | Cohort 3 (Denosumab 120 mg Q4W)
Number analyzed (Participants) | 265 | 249 | 12
Participants
  Calcium corrected Grade 3 (Above) | 0 | 1 | 0
  Calcium corrected Grade 4 (Above) | 1 | 1 | 0
  Calcium corrected Grade 3 (Below) | 1 | 0 | 0
  Calcium corrected Grade 4 (Below) | 2 | 0 | 0
  Phosphate Grade 3 (Below) | 60 | 41 | 4
  Magnesium Grade 3 (Above) | 4 | 5 | 2
  Magnesium Grade 3 (Below) | 1 | 0 | 0
  Creatinine Grade 3 (Above) | 0 | 1 | 0
  Albumin Grade 3 (Below) | 1 | 0 | 0

3. Secondary Outcome: Time to Disease Progression or Recurrence During the On-Study Period for Cohort 1, Presented as Kaplan-Meier Estimates of Probability
Description: Time to disease progression or recurrence during the on-study period was defined as the time interval (in days) from the date of first dose of study drug to the date of earliest Progressive Disease (PD) during the initial treatment phase. PD was defined as the response of progressive disease, locally recurrent disease or relapse as captured in the Disease Status page of the Case Report Form. If a participant had not had PD by the end of the initial treatment phase date, time to disease progression or recurrence were censored at her/his end of initial treatment phase date. Since median time to disease progression or recurrence for participants in cohort 1 was not reached, Kaplan-Meier estimates for the probability (expressed as a percentage) of participants in cohort 1 to have disease progression or recurrence at months 6, 12, 24, 36 and 60 are presented.
Time Frame: From first dose of study drug up to the end of the initial treatment phase (median duration approximately 30 months up to a maximum of approximately 109 months).
Population: The efficacy analysis set included all enrolled participants who were eligible for the study, and who received at least one dose of denosumab on the study. Analysis was performed on cohort 1 only.
Measure: Number (95% Confidence Interval); unit: Percent probability
Arm/Group | Cohort 1 (Denosumab 120 mg Q4W)
Number analyzed (Participants) | 260
Percent probability
  Month 6 | 1.9 [0.3 to 3.6]
  Month 12 | 4.3 [1.8 to 6.8]
  Month 24 | 6.1 [3.1 to 9.0]
  Month 36 | 8.2 [4.6 to 11.8]
  Month 60 | 11.7 [7.1 to 16.2]

4. Secondary Outcome: Percentage of Participants Without Any On-Study Surgery at Month 6 for Cohort 2
Description: The percentage of participants without any surgery at month 6 was equivalent to the number of participants without any surgery by month 6 divided by the number of cohort 2 participants who had an opportunity to complete 6 months of treatment, expressed as a percentage.
Time Frame: At month 6.
Population: The efficacy analysis set included all enrolled participants who were eligible for the study, and who received at least one dose of denosumab on the study. Analysis was performed on cohort 2 only for those who had the opportunity to be on-study for at least 6 months.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 2 (Denosumab 120 mg Q4W)
Number analyzed (Participants) | 238
Percentage of participants | 92.0 [87.8 to 95.1]

5. Secondary Outcome: Mean Serum Denosumab Trough Concentrations
Description: Blood samples for determination of serum denosumab concentration levels were obtained from participants included in the pharmacokinetic (PK) substudy at baseline (prior to administration of study drug on day 1) and at scheduled time points during the study up to week 25.
Time Frame: Blood samples were collected at baseline (day 1), days 8 and 15 and weeks 5, 9, 13 and 25.
Population: The PK analysis set included all participants who received at least 1 dose of denosumab with baseline PK measurement and at least 1 post-baseline PK measurement. Only participants with available data at each time point were included in the analysis.
Measure: Mean (Standard Deviation); unit: nanograms / milliliter
Groups:
- Adolescent PK Subset (Denosumab 120 mg Q4W): Adolescent participants enrolled in the PK substudy who received at least 1 dose of denosumab with baseline PK measurement and at least 1 post-baseline PK measurement were included in the adolescent PK analysis set. Participants received denosumab 120 mg SC Q4W, starting on study day 1, with loading doses of 120 mg SC on days 8 and 15 in the first month of treatment for those enrolled in cohorts 1 or 2.
- Adult PK Subset (Denosumab 120 mg Q4W): Adult participants enrolled in the PK substudy who received at least 1 dose of denosumab with baseline PK measurement and at least 1 post-baseline PK measurement were included in the adult PK analysis set. Participants received denosumab 120 mg SC Q4W, starting on study day 1, with loading doses of 120 mg SC on days 8 and 15 in the first month of treatment for those enrolled in cohorts 1 or 2.
Arm/Group | Adolescent PK Subset (Denosumab 120 mg Q4W) | Adult PK Subset (Denosumab 120 mg Q4W)
Number analyzed (Participants) | 10 | 15
nanograms / milliliter
  Day 1 | 0.0 (0.0) | 0.0 (0.0)
  Day 8: number analyzed (Participants) | 9 | 14
  Day 8 | 11800 (4130) | 12000 (4300)
  Day 15: number analyzed (Participants) | 9 | 13
  Day 15 | 21800 (5620) | 24200 (9050)
  Week 5: number analyzed (Participants) | 9 | 14
  Week 5 | 30400 (6150) | 33500 (8970)
  Week 9: number analyzed (Participants) | 9 | 15
  Week 9 | 25100 (6450) | 30000 (10300)
  Week 13: number analyzed (Participants) | 7 | 12
  Week 13 | 22300 (6840) | 29100 (10000)
  Week 17: number analyzed (Participants) | 7 | 13
  Week 17 | 23600 (4370) | 28300 (11600)
  Week 25: number analyzed (Participants) | 8 | 11
  Week 25 | 22400 (6690) | 25400 (10800)

ADVERSE EVENTS:
Time Frame: From first dose of study drug until last study visit; a maximum of approximately 113 months. The planned study duration for each participant was at least 60 months (following protocol amendment 7).
Description: Data are presented for the entire study duration and include AEs occurring during the treatment-emergent period (comprising both the initial treatment phase and retreatment phase) and AEs occurring after the treatment-emergent period (ie, during the safety follow-up phase).
Groups:
- Denosumab 120 mg Q4W (All Cohorts): All participants received denosumab 120 mg SC Q4W, starting on study day 1, with loading doses of 120 mg SC on days 8 and 15 in the first month of treatment for those enrolled in cohorts 1 or 2.
Arm/Group | Denosumab 120 mg Q4W (All Cohorts)
All-Cause Mortality (participants affected / at risk) | 26/526
Serious Adverse Events (participants affected / at risk) | 176/526
Other Adverse Events (participants affected / at risk) | 480/526
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Denosumab 120 mg Q4W (All Cohorts) (N=526)
Anaemia (Blood and lymphatic system disorders) | 8
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Microcytic anaemia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Bradycardia (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 2
Coronary artery disease (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Aplasia (Congenital, familial and genetic disorders) | 1
Hyperparathyroidism (Endocrine disorders) | 2
Toxic nodular goitre (Endocrine disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 2
Large intestine perforation (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Pancreatic failure (Gastrointestinal disorders) | 1
Peptic ulcer (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 2
Chest pain (General disorders) | 1
Death (General disorders) | 4
Disease recurrence (General disorders) | 1
Hernia (General disorders) | 1
Impaired healing (General disorders) | 2
Malaise (General disorders) | 1
Mucosal inflammation (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pyrexia (General disorders) | 4
Cholecystitis (Hepatobiliary disorders) | 2
Cholelithiasis (Hepatobiliary disorders) | 2
Abdominal abscess (Infections and infestations) | 1
Abdominal wall infection (Infections and infestations) | 1
Abscess (Infections and infestations) | 2
Abscess jaw (Infections and infestations) | 1
Abscess neck (Infections and infestations) | 1
Abscess oral (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 4
Arthritis infective (Infections and infestations) | 1
Aspergillus infection (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 1
Bacteroides bacteraemia (Infections and infestations) | 1
Bone abscess (Infections and infestations) | 1
Catheter site infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 2
Device related infection (Infections and infestations) | 4
Gastroenteritis (Infections and infestations) | 3
Infected cyst (Infections and infestations) | 1
Infected skin ulcer (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Infectious colitis (Infections and infestations) | 1
Muscle abscess (Infections and infestations) | 1
Orchitis (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 4
Osteomyelitis bacterial (Infections and infestations) | 1
Peritonsillar abscess (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 4
Postoperative wound infection (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Scrotal abscess (Infections and infestations) | 1
Sepsis (Infections and infestations) | 3
Staphylococcal infection (Infections and infestations) | 1
Staphylococcal osteomyelitis (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 2
Tooth infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 3
Wound infection (Infections and infestations) | 2
Wound infection staphylococcal (Infections and infestations) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Atypical femur fracture (Injury, poisoning and procedural complications) | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 3
Fracture displacement (Injury, poisoning and procedural complications) | 1
Gun shot wound (Injury, poisoning and procedural complications) | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Post procedural fistula (Injury, poisoning and procedural complications) | 1
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 1
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Pubis fracture (Injury, poisoning and procedural complications) | 1
Radiation myelopathy (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Stress fracture (Injury, poisoning and procedural complications) | 2
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 2
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Vena cava injury (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 2
Wrist fracture (Injury, poisoning and procedural complications) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 4
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Exposed bone in jaw (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 3
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 4
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 25
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bone giant cell tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 19
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bone sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ganglioneuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Myeloproliferative neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oncologic complication (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Osteosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Pelvic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rhabdomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Second primary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Spindle cell sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thyroid cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Cauda equina syndrome (Nervous system disorders) | 1
Central nervous system lesion (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Facial neuralgia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 1
Nerve compression (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 2
Spinal cord compression (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Device breakage (Product Issues) | 1
Device failure (Product Issues) | 1
Device loosening (Product Issues) | 1
Device occlusion (Product Issues) | 1
Completed suicide (Psychiatric disorders) | 1
Suicide attempt (Psychiatric disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 3
Bladder prolapse (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 2
Renal colic (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 2
Urethral fistula (Renal and urinary disorders) | 1
Urge incontinence (Renal and urinary disorders) | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal fistula (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 1
Bone lesion excision (Surgical and medical procedures) | 2
Leg amputation (Surgical and medical procedures) | 1
Spinal operation (Surgical and medical procedures) | 1
Circulatory collapse (Vascular disorders) | 1
Haematoma (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Thrombophlebitis superficial (Vascular disorders) | 1
Vasculitis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Denosumab 120 mg Q4W (All Cohorts) (N=526)
Anaemia (Blood and lymphatic system disorders) | 30
Abdominal pain (Gastrointestinal disorders) | 49
Constipation (Gastrointestinal disorders) | 60
Dental caries (Gastrointestinal disorders) | 32
Diarrhoea (Gastrointestinal disorders) | 60
Nausea (Gastrointestinal disorders) | 122
Toothache (Gastrointestinal disorders) | 68
Vomiting (Gastrointestinal disorders) | 66
Asthenia (General disorders) | 48
Fatigue (General disorders) | 142
Influenza like illness (General disorders) | 27
Oedema peripheral (General disorders) | 46
Pyrexia (General disorders) | 47
Bronchitis (Infections and infestations) | 28
Influenza (Infections and infestations) | 44
Nasopharyngitis (Infections and infestations) | 76
Upper respiratory tract infection (Infections and infestations) | 48
Procedural pain (Injury, poisoning and procedural complications) | 39
Weight increased (Investigations) | 30
Hypercalcaemia (Metabolism and nutrition disorders) | 29
Hypocalcaemia (Metabolism and nutrition disorders) | 36
Hypophosphataemia (Metabolism and nutrition disorders) | 66
Arthralgia (Musculoskeletal and connective tissue disorders) | 192
Back pain (Musculoskeletal and connective tissue disorders) | 154
Bone pain (Musculoskeletal and connective tissue disorders) | 41
Joint swelling (Musculoskeletal and connective tissue disorders) | 28
Muscle spasms (Musculoskeletal and connective tissue disorders) | 37
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 70
Myalgia (Musculoskeletal and connective tissue disorders) | 42
Neck pain (Musculoskeletal and connective tissue disorders) | 29
Pain in extremity (Musculoskeletal and connective tissue disorders) | 146
Pain in jaw (Musculoskeletal and connective tissue disorders) | 40
Dizziness (Nervous system disorders) | 34
Headache (Nervous system disorders) | 134
Hypoaesthesia (Nervous system disorders) | 38
Paraesthesia (Nervous system disorders) | 48
Anxiety (Psychiatric disorders) | 29
Depression (Psychiatric disorders) | 31
Insomnia (Psychiatric disorders) | 45
Cough (Respiratory, thoracic and mediastinal disorders) | 54
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 36
Pruritus (Skin and subcutaneous tissue disorders) | 33
Rash (Skin and subcutaneous tissue disorders) | 45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2015-09-15): https://cdn.clinicaltrials.gov/large-docs/92/NCT00680992/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-17): https://cdn.clinicaltrials.gov/large-docs/92/NCT00680992/SAP_001.pdf